CLINICAL TRIAL: NCT04224025
Title: Influence of Breath- and Movementtherapy to Clinical and Molecular Parameter in Patients With Pulmonary Hypertension
Brief Title: Training Single Arm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig, Head of centre for pulmonary hypertension, Thoraxklinik-Heidelberg gGmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Training single arm
Record Dates: First submitted 2019-12-19; First posted 2020-01-13 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Exercise; Respiratory Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise and respiratory therapy (Experimental): Rehabilitation program for three weeks in-Hospital and continuation at home
  Interventions: Other: exercise and respiratory therapy

INTERVENTIONS:
Other: exercise and respiratory therapy — three weeks in-Hospital exercise Rehabilitation program with continuation at home (total 15 weeks).

SUMMARY:
The pulmonary hypertension is a disease, which tends to a progredient right heart failure. Although there was a large progress in development of medical therapy, the quality of life, the physical efficiency and the prognosis of the patients are still limited. The aim of the study is to examine the influence of physical training to clinical and molecular parameter.

DETAILED DESCRIPTION:
The aim of this prospective, randomized, controlled study in patients with pulmonary hypertension, who are under stable optimized treatment for at least 2 months, is to examine the effect of an additional exercise and respiratory therapy.

The aim criteria measures the clinical parameters to record the effect of the training plus molecular parameter to evaluate the effectiveness of the training. The molecular parameters are composed of laboratory parameter and inflammatory parameter as well as genetic analyses, measurements of epigenetic changes measured by microRNA Expressions and DNA-methylation.

The study parameters will be assessed in the patient's routine examinations. Clinical parameters comprise of hemodynamic assessment of pulmonary arterial pressure during exercise, pump function of left and right ventricle, and further echocardiographic parameters. Improvement of exercise capacity will be measured by the change of six-minute walking distance, the breathing economics, the world health organization functional class (WHO functional class), peak oxygen consumption and blood gas analysis. The quality of life will be assessed with the SF-36 questionnaire. Data for survival analysis will be gained by structured phone interviews . The safety of the training is warranted by long-term, rest- and stress-ECG, safety laboratory, systemic blood pressure, heart frequency, oxygen saturation and occurrence of adverse events.

Patients will be examined in the Thoraxklinik Heidelberg. Patients of the training group will take part in a specific, 3-week inpatient training program at the rehabilitation center Königstuhl Heidelberg. The training program consists of exercise and respiratory therapy as well as a mental gait training. Respiratory therapy will be performed 5 times/week for 30 minutes. Furthermore, 15-25 minutes low dosed interval training on a bicycle ergometer, dumbbell training of particular muscle groups with low weights and supervised walks on ground-level will be scheduled 5-7 times/week. Three- to five times a week a "mental gait training" is conducted to estimate the patient's individual physical abilities and limitations. The heart rate during exerciseand the intensity of the training will be closely monitored and individually adjusted. After three weeks of in-hospital rehabilitation the patients are asked to continue the training for twelve further weeks at home. All patients will be examined before the training program, at the end of the in-hospital phase after three weeks and after 15 weeks.

The control examinations cover the medical history, WHO functional class, physical examination, ECG, echocardiography at rest and during exercise, spiroergometry, quality of life, blood-gas analysis, lung function, 6-minute walking distance, oxygen saturation, blood pressure and heart rate, laboratory tests. An optional magnet resonance imaging at the beginning and after three months may also be conducted. At baseline, an optional genetic assessment will be performed; and at the beginning, after three and 15 weeks the expression levels of micro RNA and methylation of the DNA will be assessed. Medication will remain stable throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Consent form
* Men and women >18 years
* Symptomatic PH (WHO-FC II-IV) invasive diagnostis with right heart catheterization: mPAP >25mmHg and a stable optimized treatment for at least 2 month
* Patients who are able to understand and agree to participate in the study

Exclusion Criteria:

* Pregnancy or breast feeding
* Variation in the medication during the last 2 months
* Patients with signs of right heart decompensation
* Major walking problems
* Unclear diagnosis
* No invasive clarification of the PH
* Acute illness, infections and fever
* Grave lung disease with FEV1 <50% or TLC <70% from target
* Further conclusion criteria are followed: acrive myokarditis, unstable angina pectoris, movement induced ventricular rhythmdisturbance, decompensation of the right hart insufficiency, meaningful heartvitien, hyperthrophic obstructive cardiomyopathie or a high grade reduced left ventricular pump function
* Acute psychosis or other conditions which appears a reduced understanding
* Patiets with metallic valvular or other metallic implants
* Incorporated ferromagnetic materials or for the MRI incompatibel activce medicinal products
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-11-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
6-minute Walking distance | change from baseline to final assessment after 3 months
  Walking distance in metres

SECONDARY OUTCOMES:
Peak oxygen consumption | change from baseline to final assessment after 3 months
  Peak oxygen consumption during cardiopulmonary exercise testing
Ventilatory equivalent, assessed during cardiopulmonary exercise testing at Peak exercise | change from baseline to final assessment after 3 months
  Ventilatory equivalent during cardiopulmonary exercise testing
Workload during cardiopulmonary exercise testing | change from baseline to final assessment after 3 months
  Peak workload in Watts
Epigenetic mechanisms; changes in micro RNA methylation/expression | change from baseline to final assessment after 3 months
  changes in epigenetic mechanisms
Echocardiography systolic pulmonary arterial pressure | change from baseline to final assessment after 3 months
  systolic pulmonary arterial pressure
Echocardiography right ventricular area | change from baseline to final assessment after 3 months
  right ventricular area in cm^2
Echocardiography right atrial area | change from baseline to final assessment after 3 months
  right atrial area in cm^2
Echocardiography tricuspid annular plane systolic excursion | change from baseline to final assessment after 3 months
  tricuspid annular plane systolic excursion
Echocardiography right ventricular pump function | change from baseline to final assessment after 3 months
  right ventricular pump function qualitative
World Health Organization functional class | change from baseline to final assessment after 3 months
  functional class of patient's symptoms
Laboratory NT-proBNP | change from baseline to final assessment after 3 months
  NT-proBNP as marker of right heart insufficiency
Quality of life physical Summation score; scores from 0-100 with higher scores indicating better outcome | change from baseline to final assessment after 3 months
  short form health Survey 36 physical Summation score
Quality of life mental Summation score; scores from 0-100 with higher scores indicating better outcome | change from baseline to final assessment after 3 months
  short form health Survey 36 mental Summation score
Blood gas Analysis Oxygen saturation | change from baseline to final assessment after 3 months
  Oxygen Saturation at rest

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Pulmonary Hypertension at the Thoraxklinik, Heidelberg University Hospital, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes